CLINICAL TRIAL: NCT01613248
Title: A Phase IIb, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study of MK-1602 in the Treatment of Acute Migraine
Brief Title: A Dose-Finding Study of MK-1602 in the Treatment of Acute Migraine (MK-1602-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1602-006
Record Dates: First submitted 2012-05-16; First posted 2012-06-07 (Estimated); Results first posted 2016-09-30 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- MK-1602 1 mg (Experimental): MK-1602 1 mg single dose as treatment for a moderate or severe migraine headache. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 10 mg (Experimental): MK-1602 10 mg single dose as treatment for a moderate or severe migraine headache. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 25 mg (Experimental): MK-1602 25 mg single dose as treatment for a moderate or severe migraine headache. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 50 mg (Experimental): MK-1602 50 mg single dose as treatment for a moderate or severe migraine headache. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 100 mg (Experimental): MK-1602 100 mg single dose as treatment for a moderate or severe migraine headache. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- Placebo (Placebo Comparator): Placebo-matching MK-1602 single dose as treatment for a moderate or severe migraine headache. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: Placebo-matching MK-1602; Drug: Rescue medication

INTERVENTIONS:
Drug: MK-1602 — Single 1, 10, 25, 50 or 100 mg dose of MK-1602 taken at onset of migraine of moderate or severe intensity. Dosage form is film coated tablet for oral administration. Dose is provided to participants as a blinded bottle of tablets packaged to achieve the various MK-1602 dose levels to be studied. Participants will be instructed to take all study medication from the bottle when they treat their migraine headache.
  Arms: MK-1602 1 mg; MK-1602 10 mg; MK-1602 100 mg; MK-1602 25 mg; MK-1602 50 mg
Drug: Placebo-matching MK-1602 — Single administration of placebo-matching MK-1602 taken at onset of migraine of moderate or severe intensity. Dosage form is film coated tablet for oral administration. Dose is provided to participants as a blinded bottle of tablets packaged to achieve placebo study medication. Participants will be instructed to take all study medication from the bottle when they treat their migraine headache.
  Arms: Placebo
Drug: Rescue medication — If moderate or severe migraine headache pain continues 2 hours after dose of study medication or if migraine headache comes back within 48 hours,
  Participants will be allowed to take their own rescue migraine medication, which may include analgesics (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs]), anti-emetics, triptans or other medication not explicitly excluded.

SUMMARY:
The purpose of this study is to assess the effectiveness, safety and tolerability of a range of doses of MK-1602 versus placebo in the treatment of acute migraine.

ELIGIBILITY:
Inclusion Criteria:

* > 1 year history of migraine with or without aura as defined by International Headache Society (IHS) criteria 1.1 and/or 1.2
* Migraines typically last between 4 to 72 hours, if untreated
* ≥ 2 and ≤ 8 moderate or severe migraine attacks per month in each of

the two months prior to screening

* Male, female who is not of reproductive potential, or female of

reproductive potential with a screening serum β-human chorionic gonadotropin (β-hCG) level consistent with a not-pregnant state, and who agrees to use acceptable contraception

Exclusion Criteria:

* Pregnant or breast-feeding, or is a female expecting to conceive within the projected duration of study participation
* Participant has difficulty distinguishing his/her migraine attacks from tension-type headaches
* History of predominantly mild migraine attacks or migraines that usually

resolve spontaneously in less than two hours

* More than 15 headache-days per month or has taken medication for acute headache on more than 10 days per month in any of the three months prior to screening
* Basilar-type or hemiplegic migraine headache
* > 50 years old at age of migraine onset
* Taking migraine prophylactic medication where the prescribed daily dose

has changed during the 3 months prior to screening and will not be changed

during the study

* Taking a proton pump inhibitor (PPI) or a histamine receptor 2 (H2) blocker on a daily or near daily basis (> 3 days per week)
* Taking the following medications from 1 month prior to screening through study period: potent cytochrome P450 (CYP) 3A4 inhibitors (e.g., cyclosporine, itraconazole, ketoconazole, fluconazole, erythromycin, clarithromycin, nefazodone, telithromycin, cimetidine, quinine, diltiazem, verapamil, and human immunodeficiency virus [HIV] protease inhibitors), moderate or marked CYP3A4 inducers (e.g., rifampicin, rifabutin, barbiturates [e.g., phenobarbital and primidone], systemic glucocorticoids, nevirapine, efavirenz, pioglitazone, carbamazepine, phenytoin, and St. Johns wort), or drugs with narrow therapeutic margins and potential for drug interactions in the CYP2C family (e.g., warfarin)
* Participant is unable to refrain from consumption of grapefruit or grapefruit juice during study
* History of hypersensitivity to, or has experienced a serious adverse event

in response to 3 or more classes of drugs (prescription and over-the-counter)

* Clinical or laboratory evidence of uncontrolled diabetes, human immunodeficiency virus (HIV) disease, or significant pulmonary, renal, hepatic, endocrine, or other systemic disease
* Other confounding pain syndromes, psychiatric conditions such as uncontrolled major depression, dementia or significant neurological disorders other than migraine. Patients who are currently being treated with non-prohibited medication for depression and symptoms are well controlled are eligible to participate
* Participant is at imminent risk of self-harm
* History of malignancy ≤ 5 years prior to study, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* History of gastric or small intestinal surgery (including gastric bypass

surgery or banding), or presence of a disease that causes malabsorption

* Participant has recent history (within the last year) of drug or alcohol abuse or dependence or is a user of recreational or illicit drugs
* Participant is legally or mentally incapacitated
* Donation of blood products or phlebotomy of > 300 ml within 8

weeks of study, or intent to donate blood products or receive

blood products within 30 days of screening and throughout study

* Intent to donate eggs or sperm within the projected duration of the

study

* Current participation in or participation within 30 days of screening

in a study with an investigational compound or device

* Previous exposure to MK-0974 and/or MK-3207
* Use within the past 2 months of an opioid- or barbiturate-containing

analgesic for migraine relief

* Inpatient or emergency department treatment of an acute migraine

attack within the past 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

REFERENCES:
- [Background] Voss T, Lipton RB, Dodick DW, Dupre N, Ge JY, Bachman R, Assaid C, Aurora SK, Michelson D. A phase IIb randomized, double-blind, placebo-controlled trial of ubrogepant for the acute treatment of migraine. Cephalalgia. 2016 Aug;36(9):887-98. doi: 10.1177/0333102416653233. Epub 2016 Jun 6. PMID 27269043
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Started | 139 | 138 | 139 | 139 | 139 | 140
Completed | 110 | 104 | 106 | 101 | 104 | 102
Not Completed | 29 | 34 | 33 | 38 | 35 | 38
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 5 | 0 | 1
Not completed — Lost to Follow-up | 5 | 7 | 4 | 8 | 4 | 2
Not completed — Study Terminated by Sponsor | 4 | 6 | 8 | 8 | 9 | 11
Not completed — Physician Decision | 8 | 8 | 9 | 4 | 7 | 6
Not completed — Lack of Qualifying Event | 9 | 11 | 10 | 11 | 15 | 18
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Subjects as Treated Population included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg | Total
Number analyzed (Participants) | 113 | 107 | 108 | 104 | 106 | 102 | 640
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (11.7) | 39.6 (10.7) | 41.1 (10.9) | 41.4 (11.5) | 40.7 (12.3) | 41.9 (11.0) | 40.8 (11.4)
Age, Customized [Number; unit: participants]
  < 20 years | 1 | 1 | 0 | 2 | 2 | 0 | 6
  20 to 29 years | 18 | 21 | 19 | 13 | 19 | 16 | 106
  30 to 39 years | 42 | 29 | 28 | 32 | 32 | 26 | 189
  40 to 49 years | 22 | 36 | 42 | 33 | 23 | 33 | 189
  50 to 59 years | 19 | 17 | 14 | 16 | 21 | 23 | 110
  60 to 64 years | 10 | 2 | 5 | 8 | 9 | 3 | 37
  >= 65 years | 1 | 1 | 0 | 0 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 95 | 92 | 91 | 92 | 90 | 559
  Male | 14 | 12 | 16 | 13 | 14 | 12 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Pain Freedom (PF) at 2 Hours Post-Dose
Description: PF was defined as a reduction in headache severity from Grade 2 or 3 at Baseline to Grade 0. Headache severity was reported by the participant using a 4-point scale where: 0=no pain, 1=mild pain, 2=moderate pain and 3=severe pain.
Time Frame: 2 hours post-dose
Population: Participants from the Full Analysis Set, all participants who received treatment and had both a Baseline and at least one post-dose efficacy measurement, with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 112 | 107 | 108 | 103 | 105 | 102
percentage of participants | 8.9 [4.4 to 15.8] | 5.6 [2.1 to 11.8] | 14.8 [8.7 to 22.9] | 21.4 [13.9 to 30.5] | 21.0 [13.6 to 30.0] | 25.5 [17.4 to 35.1]

2. Primary Outcome: Percentage of Participants Reporting Pain Relief (PR) at 2 Hours Post-Dose
Description: PR was defined as a reduction of a moderate or severe migraine headache (Grade 2 or 3) at Baseline to a mild headache or no headache (Grade 1 or 0) 2 hours post-dose. Headache severity was reported by the participant using a 4-point scale where: 0=no pain, 1=mild pain, 2=moderate pain and 3=severe pain.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 112 | 107 | 108 | 103 | 105 | 102
percentage of participants | 44.6 [35.2 to 54.3] | 37.4 [28.2 to 47.3] | 52.8 [42.9 to 62.5] | 53.4 [43.3 to 63.3] | 57.1 [47.1 to 66.8] | 58.8 [48.6 to 68.5]

3. Primary Outcome: Number of Participants With One or More Adverse Events Within 48 Hours Post-Dose
Description: An AE is any unfavorable and unintended change in the structure (signs), function (symptoms), or chemistry (laboratory data) of the body temporally associated with any use of a sponsor product, whether or not considered related to the use of the product.
Time Frame: Up to 48 hours post-dose
Population: All Subjects as Treated (ASaT) population included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 103 | 107 | 102
participants | 28 | 33 | 29 | 21 | 23 | 30

4. Primary Outcome: Number of Participants With One or More Adverse Events Within 14 Days Post-Dose
Description: as for outcome 3
Time Frame: Up to 14 days post-dose
Population: ASaT population included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 103 | 107 | 102
participants | 33 | 37 | 32 | 24 | 30 | 32

5. Primary Outcome: Number of Participants Who Discontinued From Study Due to Adverse Events
Time Frame: Up to 5 weeks post-dose
Population: ASaT population included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 104 | 106 | 102
participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Reporting Absence of Phonophobia at 2 Hours Post-Dose
Description: Phonophobia is sensitivity to loud sounds.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 112 | 107 | 108 | 103 | 105 | 102
percentage of participants | 42.0 [32.7 to 51.7] | 45.8 [36.1 to 55.7] | 49.1 [39.3 to 58.9] | 55.3 [45.2 to 65.1] | 56.2 [46.2 to 65.9] | 60.8 [50.6 to 70.3]

7. Secondary Outcome: Percentage of Participant Reporting Absence of Photophobia at 2 Hours Post-Dose
Description: Photophobia is sensitivity to bright light.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 112 | 107 | 108 | 103 | 105 | 102
percentage of participants | 30.4 [22.0 to 39.8] | 37.4 [28.2 to 47.3] | 43.5 [34.0 to 53.4] | 39.8 [30.3 to 49.9] | 47.6 [37.8 to 57.6] | 54.9 [44.7 to 64.8]

8. Secondary Outcome: Percentage of Participants Reporting Absence of Nausea at 2 Hours Post-Dose
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 112 | 107 | 108 | 103 | 105 | 102
percentage of participants | 62.5 [52.9 to 71.5] | 59.8 [49.9 to 69.2] | 67.6 [57.9 to 76.3] | 73.8 [64.2 to 82.0] | 68.6 [58.8 to 77.3] | 70.6 [60.7 to 79.2]

9. Secondary Outcome: Percentage of Participants Reporting Sustained Pain Freedom (SPF) 2-24 Hours Post-Dose
Description: SPF was defined as PF at 2 hours post-dose, with no administration of any rescue medication and with no occurrence of a mild/moderate/severe headache during the 24 hour period after dosing with study medication.
Time Frame: 2-24 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 103 | 106 | 102
percentage of participants | 6.2 [2.5 to 12.3] | 4.7 [1.5 to 10.6] | 9.3 [4.5 to 16.4] | 14.6 [8.4 to 22.9] | 15.1 [8.9 to 23.4] | 21.6 [14.0 to 30.8]

10. Secondary Outcome: Percentage of Participants Reporting SPF 2-48 Hours Post-Dose
Description: SPF was defined as PF at 2 hours post-dose, with no administration of any rescue medication and with no occurrence of a mild/moderate/severe headache during the 48 hour period after dosing with study medication.
Time Frame: 2-48 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 103 | 106 | 102
percentage of participants | 6.2 [2.5 to 12.3] | 4.7 [1.5 to 10.6] | 9.3 [4.5 to 16.4] | 14.6 [8.4 to 22.9] | 14.2 [8.1 to 22.3] | 20.6 [13.2 to 29.7]

11. Secondary Outcome: Percentage of Participants Reporting Sustained Pain Relief (SPR) 2-24 Hours Post-Dose
Description: SPR was defined as PR at 2 hours post-dose, with no administration of any rescue medication and with no occurrence of a moderate/severe headache during the 24 hour period after dosing with study medication.
Time Frame: 2-24 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 103 | 105 | 102
percentage of participants | 28.3 [20.2 to 37.6] | 17.8 [11.0 to 26.3] | 36.1 [27.1 to 45.9] | 39.8 [30.3 to 49.9] | 45.7 [36.0 to 55.7] | 46.1 [36.2 to 56.2]

12. Secondary Outcome: Percentage of Participants Reporting SPR 2-48 Hours Post-Dose
Description: SPR was defined as PR at 2 hours post-dose, with no administration of any rescue medication and with no occurrence of a moderate/severe headache during the 48 hour period after dosing with study medication.
Time Frame: 2-48 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 112 | 106 | 108 | 103 | 105 | 102
percentage of participants | 25.0 [17.3 to 34.1] | 17.0 [10.4 to 25.5] | 32.4 [23.7 to 42.1] | 37.9 [28.5 to 48.0] | 42.9 [33.2 to 52.9] | 43.1 [33.4 to 53.3]

13. Secondary Outcome: Percentage of Participants Reporting Total Migraine Freedom (TMF) at 2 Hours Post-Dose
Description: TMF at 2 hours post dose was defined as PF with no photophobia, phonophobia, nausea, or vomiting at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 112 | 107 | 108 | 103 | 105 | 102
percentage of participants | 8.0 [3.7 to 14.7] | 5.6 [2.1 to 11.8] | 13.9 [8.0 to 21.9] | 20.4 [13.1 to 29.5] | 20.0 [12.8 to 28.9] | 23.5 [15.7 to 33.0]

14. Secondary Outcome: Percentage of Participants Reporting TMF at 2-24 Hours Post-Dose
Description: TMF at 2-24 hours post-dose was defined as SPF with no photophobia, phonophobia, nausea, or vomiting during the 2 to 24 hour period after dosing with study medication.
Time Frame: 2-24 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 103 | 106 | 102
percentage of participants | 5.3 [2.0 to 11.2] | 4.7 [1.5 to 10.6] | 9.3 [4.5 to 16.4] | 12.6 [6.9 to 20.6] | 14.2 [8.1 to 22.3] | 20.6 [13.2 to 29.7]

15. Secondary Outcome: Percentage of Participants Reporting TMF at 2-48 Hours Post-Dose
Description: TMF at 2-48 hours post-dose was defined as SPF with no photophobia, phonophobia, nausea, or vomiting during the 2 to 48 hour period after dosing with study medication.
Time Frame: 2-48 hours post-dose
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 113 | 107 | 108 | 103 | 106 | 102
percentage of participants | 5.3 [2.0 to 11.2] | 4.7 [1.5 to 10.6] | 9.3 [4.5 to 16.4] | 12.6 [6.9 to 20.6] | 13.2 [7.4 to 21.2] | 19.6 [12.4 to 28.6]

ADVERSE EVENTS:
Description: All Subjects as Treated Population, all randomized participants who received at least 1 dose of study treatment, was used to determine the number of participants at risk for Serious Adverse Events (SAE) and Other Adverse Events.
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/107 | 0/108 | 0/104 | 1/106 | 0/102
Other Adverse Events (participants affected / at risk) | 15/113 | 22/107 | 13/108 | 15/104 | 14/106 | 17/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=113) | MK-1602 1 mg (N=107) | MK-1602 10 mg (N=108) | MK-1602 25 mg (N=104) | MK-1602 50 mg (N=106) | MK-1602 100 mg (N=102)
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 — SAE: Myoclonus occurred 15 days post-dose.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=113) | MK-1602 1 mg (N=107) | MK-1602 10 mg (N=108) | MK-1602 25 mg (N=104) | MK-1602 50 mg (N=106) | MK-1602 100 mg (N=102)
Dry mouth (Gastrointestinal disorders) | 4 | 8 | 2 | 3 | 4 | 5
Nausea (Gastrointestinal disorders) | 4 | 7 | 4 | 6 | 8 | 7
Dizziness (Nervous system disorders) | 1 | 8 | 5 | 3 | 2 | 6
Somnolence (Nervous system disorders) | 6 | 5 | 4 | 5 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.